CLINICAL TRIAL: NCT05755269
Title: Genetic Risk Estimation in Breast Cancer and Assessing Health Disparities
Brief Title: Adding a Genetic Risk Evaluation to Standard Breast Cancer Risk Assessment for African American and Hispanic Women
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC220303; NCI-2022-10133 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-003513 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2023-02-14; First posted 2023-03-06 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Breast Atypical Ductal Hyperplasia; Breast Atypical Lobular Hyperplasia; Breast Carcinoma; Breast Lobular Carcinoma In Situ
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms; Breast Carcinoma In Situ | interventions — Specimen Handling; Genotype

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (blood collection, genotyping, surveys): Patients complete a survey and undergo collection of a blood sample for PRS genotyping at baseline. Patients receive their PRS results and complete another survey 6 weeks to 6 months after baseline and then complete surveys annually over 10 years on study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Genotyping; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Genotyping — Undergo genotyping
  Other Names: GENOTYPE; Genotype Analysis; Genotype Assay
Other: Survey Administration — Complete surveys

SUMMARY:
This study evaluates whether adding a polygenic risk score evaluation to standard breast cancer risk assessment tools helps African American and Hispanic women make more informed decisions about accepting additional breast cancer screening and prevention strategies. Traditional breast cancer risk assessments rely mostly on the presence of standard clinical risk factors including family history, reproductive history, and mammographic breast density. This information can be combined with validated risk estimation models to provide a measure of a patient's 10 year and lifetime risk for breast cancer. A polygenic risk score helps to estimate breast cancer risk in a more individualized way by evaluating a patient's genetics. Adding a polygenic risk score evaluation to traditional screening techniques may help minority women make more informed decisions about screening and prevention strategies for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To explore if the addition of an individual polygenic risk score (PRS) to the Breast Cancer Risk Assessment Tool (BCRAT) or Tyrer-Cuzick (IBIS) score will improve intentions to adhere to recommended breast cancer screening strategies such as mammography, magnetic resonance imaging (MRI), or molecular breast Imaging in women of underserved racial minorities.

II. To explore if the addition of the PRS to the BCRAT or IBIS risk score will aid women in deciding whether to take preventative endocrine therapy in women of racial minorities.

III. To understand how individualized risk assessment and information on PRS may alter perceived risk of breast cancer.

IV. To follow this cohort of women over 10 years to determine subsequent outcomes in regards to diagnoses of at-risk lesions or cancer.

OUTLINE: This is an observational study.

Patients complete a survey and undergo collection of a blood sample for PRS genotyping at baseline. Patients receive their PRS results and complete another survey 6 weeks to 6 months after baseline and then complete surveys annually over 10 years on study.

ELIGIBILITY:
Inclusion Criteria:

* Women who self-identify as African American/Black or Hispanic/Latinx
* Women >= 30 years old and =< 75 years old
* Women with any of the following:

  * IBIS (Tyrer-Cuzik) score of >= 5% for the 10 year risk OR
  * BCRAT (Gail Model) score of > 3 % for the 5 year risk
  * History of biopsy proven atypical ductal hyperplasia or atypical lobular hyperplasia (with risk calculator assessment A and B)
  * History of biopsy proven lobular carcinoma in situ (with risk calculator assessment A and B)
* Able to participate in all aspects of the study
* Understand and signed the study informed consent

Exclusion Criteria:

* Women whose calculated risk for breast cancer falls below the threshold
* Unable to give informed consent
* Prior history of invasive breast cancer, ductal carcinoma in situ or other breast cancers
* Women who are pregnant or breastfeeding
* Prior use of prevention drugs for longer than 6 months
* Prior risk reducing or prophylactic mastectomy
* Known pathogenic genetic mutation linked to breast cancer (such as BRCA 1/2, PALB2, ATM, CHEK2)

Ages: 30 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: African American/Black or Hispanic/Latinx women attending the Mayo Clinic Breast Center.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2033-01-15 (Estimated); Study Completion 2033-01-15 (Estimated)

PRIMARY OUTCOMES:
Whether the addition of an individual polygenic risk score (PRS) to the Breast Cancer Risk Assessment Tool (BCRAT) will improve intentions to adhere to recommended breast cancer screening strategies | Up to 10 years
  Continuous variables will be summarized as mean (standard deviation) or median (range) and categorical variables will be reported as frequency (percentage).
Whether the addition of an individual polygenic risk score (PRS) to the Tyrer-Cuzick (IBIS) score will improve intentions to adhere to recommended breast cancer screening strategies | Up to 10 years
  Continuous variables will be summarized as mean (standard deviation) or median (range) and categorical variables will be reported as frequency (percentage).
Whether the addition of the PRS to the BCRAT will aid women in deciding whether to take preventative endocrine therapy in women of racial minorities | Up to 10 years
  PRS score will be generated using a statistical model to determine a woman's absolute risk of breast cancer, by adding the PRS to the predictions based on either the BCRAT or IBIS models. Continuous variables will be summarized as mean (standard deviation) or median (range) and categorical variables will be reported as frequency (percentage).
Whether the addition of the PRS to the IBIS risk score will aid women in deciding whether to take preventative endocrine therapy in women of racial minorities | Up to 10 years
  PRS score will be generated using a statistical model to determine a woman's absolute risk of breast cancer, by adding the PRS to the predictions based on either the BCRAT or IBIS models. Continuous variables will be summarized as mean (standard deviation) or median (range) and categorical variables will be reported as frequency (percentage).
How individualized risk assessment on PRS may alter perceived risk of breast cancer | Up to 10 years
  PRS score will be generated using a statistical model to determine a woman's absolute risk of breast cancer, by adding the PRS to the predictions based on either the BCRAT or IBIS models. Will use the R package Individualized Coherent Absolute Risk Estimators (iCare) a tool that allows researchers to quickly build models for absolute risk and apply them to estimate individuals' risk based on a set of user defined input. Continuous variables will be summarized as mean (standard deviation) or median (range) and categorical variables will be reported as frequency (percentage).
How individualized information on PRS may alter perceived risk of breast cancer | Up to 10 years
  The information used to calculate risk based on either the BCRAT or IBIS models accounts for known risk factors other than the PRS, creating a baseline hazard rate for each woman. Continuous variables will be summarized as mean (standard deviation) or median (range) and categorical variables will be reported as frequency (percentage).
Long-term cumulative risk of cancer for the at-risk lesion | Up to 10 years
  Kaplan-Meier method will be used to estimate the long-term cumulative risk of cancer for the at-risk lesion.

CONTACTS AND LOCATIONS:
Overall Officials: Sabrina Sahni, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials